CLINICAL TRIAL: NCT01678664
Title: Everolimus as Treatment After Embolization or Chemoembolization for Liver Metastases From Digestive Endocrine Tumors
Brief Title: Everolimus After (Chemo)Embolization for Liver Metastases From Digestive Endocrine Tumors
Acronym: EVACEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFCD 1104
Record Dates: First submitted 2012-08-22; First posted 2012-09-05 (Estimated); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Neuroendocrine Tumors; Hepatic Metastases; Metastases
Keywords: cancer; neuroendocrine tumors; gastrointestinal tract; metastases; liver; hepatic
MeSH Terms: conditions — Neuroendocrine Tumors; Neoplasm Metastasis; Neoplasms | interventions — Everolimus; Embolization, Therapeutic; Doxorubicin; Chemoembolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- embolization or chemoembolization plus everolimus (Experimental): After 2 sessions of embolization with microsphere of 100 to 500 µm or chemoembolization with 100 mg of doxorubicine and 10 ml of lipiodol, administered every day, 10 mg of everolimus during 24 months or until progression (hepatic and other site).
  Interventions: Drug: Everolimus; Device: embolization; Drug: Doxorubicin

INTERVENTIONS:
Drug: Everolimus — 10 mg per day of everolimus during 24 months or until progression disease
Device: embolization — 2 sessions embolization with spheric particles
  Other Names: spheric particules of 100 to 500 µm
Drug: Doxorubicin — 2 sessions chemoembolization with 10 mg of lipiodol with 100 mg of doxorubicine
  Other Names: Chemoembolization

SUMMARY:
Determine wether 24 months treatment with everolimus prolongs progression free survival rate (based on a central assessment) after embolisation ou chemoembolisation for liver metastases.

* H0 a 24 months progression free survival rate less than 35% is unacceptable
* H1 a 24 months progression free survival rate greater than 35% would show that everolimus treatment is beneficial, the expected 24 months progression free survival rate being 50%

ELIGIBILITY:
Inclusion Criteria:

* Well differentiated (grade 1 and 2 according to WHO classification 2010 appendix 2), histologically-proven endocrine tumor of the gastrointestinal tract (TENpath review mandatory),
* Measurable liver metastasis (or metastases) as defined in RECIST v1.1 that are unresectable and inaccessible to radiofrequency ablation-type local treatment
* Hepatic arterial embolization or chemoembolization indicated for tumor size reduction, confirmed in an multidisciplinary team (MDT) meeting, due to the progressive nature of the liver metastases (morphological progression during the past 12 months as defined in RECIST v1.1)
* Age ≥ 18 years
* WHO performance status ≤ 2
* No contraindications to embolization or chemoembolization or everolimus
* Satisfactory laboratory assessments:Neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, Hb > 10 g/dL, serum bilirubin ≤ 1.5 x the upper limit of normal (ULN), INR < 1.3 (or < 3 for patients on anticoagulant therapy) ALT and AST ≤ 5 x ULN, creatinine ≤ 1.5 x ULN, fasting serum cholesterol ≤ 300 mg/dL or 7.75 mmol/L and triglycerides ≤ 2.5 x ULN (if either or both of these limits are exceeded, the patient may only be included into the study after institution of appropriate lipid-lowering therapy)
* Complete resolution of toxic effects of any prior treatments, or persistence at grade 1 at most (CTCAE version 4.0)
* Minimum time since previous treatment: 28 days
* Patient has been informed and has signed an informed consent form, after verification of the eligibility criteria
* Patient covered by a French national health insurance scheme

Exclusion Criteria:

* Duodenopancreatic neuroendocrine tumor
* Poorly differentiated and/or grade 3 endocrine tumor,
* Embolization or chemoembolization indicated for symptomatic control only
* Prior hepatic TACE or embolization
* Prior treatment with an mTOR inhibitor (somatostatin analogs to control secretion are permitted)
* Symptomatic bone metastasis (or metastases)
* Any uncontrolled progressive disease: hepatic failure, renal failure, respiratory failure, NYHA class III-IV congestive heart failure, unstable angina, myocardial infarction, significant arrhythmia
* Interstitial lung disease
* Uncontrolled diabetes, defined by HbA1c > 8%
* Chronic corticosteroid or immunosuppressant therapy
* Hypersensitivity to everolimus, other rapamycin derivatives, or one of the excipients
* Major surgery, open biopsy, or significant traumatic lesion during the 28 days prior to starting the investigational treatment Incompletely healed wound or foreseeable need for major surgery during the study
* Contraindication to vascular occlusion procedures: Portal thrombosis, biliodigestive anastomosis
* Malignancy during the past 5 years, with the exception of curatively treated basal cell skin carcinoma or in situ cervical cancer
* Foreseeable non-compliance
* Medical, geographic, sociological, psychological, or legal situation that would preclude the patient from completing the study or signing an informed consent form
* Pregnant or breast-feeding women
* Men or women of child-bearing potential not using effective contraception
* Concurrent participation in another investigational study that could affect the primary endpoint of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas WALTER, PhD, Principal Investigator — Hôpital Edouard Herriot - Lyon
Locations (18):
- France (18):
  - CHU - Hôtel Dieu, Angers
  - Hôpital Avicenne, Bobigny
  - Hôpital Saint André, Bordeaux
  - Hôpital Côte de Nacre, Caen
  - CHU - Estaing, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - Centre GF Leclerc, Dijon
  - CHU - Hôpital François Mitterand, Dijon
  - Hôpital Edouard Herriot, Lyon
  - CHU La Timone, Marseille
  - CHR, Orléans
  - CHU Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Robert Debré, Reims
  - CHU, Rouen
  - Hôpital Rangueil, Toulouse
  - Hôpital Trousseau, Tours
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Walter T, Lepage C, Coriat R, Barbier E, Cadiot G, Caroli-Bosc FX, Aparicio T, Bouhier-Leporrier K, Hentic-Dhome O, Gay F, Dupont-Gossart AC, Duluc M, Lepere C, Lecomte T, Smith D, Petorin C, Di-Fiore F, Ghiringhelli F, Legoux JL, Guimbaud R, Baudin E, Lombard-Bohas C, de Baere T; FFCD 1104 investigators/investigators. Everolimus after hepatic arterial embolisation therapy of metastases from gastrointestinal neuroendocrine tumours: The FFCD 1104-EVACEL-GTE phase II study. Eur J Cancer. 2019 Dec;123:92-100. doi: 10.1016/j.ejca.2019.09.021. Epub 2019 Oct 31. PMID 31678771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 28th December 2012 and 16t March 2016, 74 patients were included by 19 french centers. Actual start date was actulaized in the protocol section.
Pre-assignment Details: Before enrollement, standard examinations (biological, clinical) were done. In terms of imaging, abdominal and thoracic computed tomography scan or MRI were also done.
Period: Overall Study
Arm/Group | Embolization or Chemoembolization Plus Everolimus
Started | 74
Completed | 74
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All the patients enrolled in the study
Arm/Group | Embolization or Chemoembolization Plus Everolimus
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 74
Region of Enrollment [Number; unit: participants]
  France | 74

OUTCOME MEASURES:

1. Primary Outcome: Rate of Hepatic Progression Free Survival at 24 Months
Description: Hepatic progression free survival rate as defined in RECIST 1.1 (with death considered as progression) during the 24 months of treatment with everolimus.
  Progression-free survival rate (PFS) (based on the investigator) according to RECIST v1.1 according to RECIST v1.1 will be defined as the time from the date of inclusion to the date of hepatic progression or death (due to any cause). For patients who are alive with no hepatic progression, it will be defines as the time from the date of inclusion and the date of the last tumor assessment.
Time Frame: Up to 24 months
Population: The analysis population for the primary endpoint was defined as the population of evaluable patients. A patient was considered evaluable if he or she hadreceived at least one dose of everolimus and at least one image on treatment.
  A patient who died (from any cause after treatment) or progressed to liver disease before 24 months was evaluable and considered a failure for the primary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Embolization or Chemoembolization Plus Everolimus
Number analyzed (Participants) | 67
Participants
  Patients with hepatic progression or DCD at 24 months | 47
  Patients alive without hepatic progression at 24 months | 20

2. Secondary Outcome: Progression-free Survival (Hepatic or Not)
Description: Progression-free survival rate was defined as the time from the date of inclusion to the date of disease progression (hepatic or not) evaluated by RECIST V1.1 criteria or death (due to any cause) or the date of the last news for alive patients
Time Frame: From randomization until the date of first progression (clinical or radiological) or death from any cause whichever came first, assessed up to 3 years
Population: All patients included in the study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Embolization or Chemoembolization Plus Everolimus
Number analyzed (Participants) | 74
months | 16.9 [12.6 to 22.4]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of inclusion to the date of death, regardless of the cause of death, or the date of last contact for patients who are alive.
Time Frame: From randomization until death or last news for alive patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Embolization or Chemoembolization Plus Everolimus
Number analyzed (Participants) | 74
Months | 51.0 [33.0 to 60.3]

ADVERSE EVENTS:
Time Frame: Up to the end of treatment Death were monitored even the patient has stopped the study treatment (up to 5 years) whereas adverse events were monitored until the end of the study protocol (average of treatment=24 months)
Arm/Group | Embolization or Chemoembolization Plus Everolimus
All-Cause Mortality (participants affected / at risk) | 32/74
Serious Adverse Events (participants affected / at risk) | 35/74
Other Adverse Events (participants affected / at risk) | 67/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Embolization or Chemoembolization Plus Everolimus (N=74)
Anaemia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 2
Cardiac Failure (Cardiac disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
General physical health deterioration (General disorders) | 6
Hyperthermia (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 5
Cholecystitis acute (Hepatobiliary disorders) | 2
Sepsis (Infections and infestations) | 2
Malnutrition (Metabolism and nutrition disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Embolization or Chemoembolization Plus Everolimus (N=74)
Fatigue (General disorders) | 59
Fever (General disorders) | 25
Infections (Infections and infestations) | 21
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Peripheral Oedema (General disorders) | 26
Deep Thrombosis (Vascular disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 61
Leukopenia (Blood and lymphatic system disorders) | 38
Neutropenia (Blood and lymphatic system disorders) | 21
Lymphopenia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 35
Dysguesia (Gastrointestinal disorders) | 8
Mucositis/stomatitis (Gastrointestinal disorders) | 32
Weight loss (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 47
Abdominal pain (Gastrointestinal disorders) | 27
Anorexia (Gastrointestinal disorders) | 21
Nausea (Gastrointestinal disorders) | 25
Vomiting (Gastrointestinal disorders) | 22
Dry Skin (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 7
Nail disorders (Skin and subcutaneous tissue disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15
Biological liver toxicity (Investigations) | 64
Hypercholesterolemia (Investigations) | 37
Hypertriglyceridemia (Investigations) | 38
Hyperglycaemia (Investigations) | 51
Hypoalbuminumia (Investigations) | 11
Hypocalcemia (Investigations) | 26
Hypokalaemia (Investigations) | 11
Hyponatraemia (Investigations) | 23
Hypomagnesaemia (Investigations) | 14
Hypophosphataemia (Investigations) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-08-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT01678664/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT01678664/SAP_001.pdf